CLINICAL TRIAL: NCT06685939
Title: To Investigate The Difference of Complications and Short-term Prognosis Between Laparoscopic and Open Pancreaticoduodenectomy in Patients With Pancreatic Cancer Based on a Special Disease Cohort Database
Brief Title: The Differences of Complications Between LPD(Laparoscopic Pancreaticoduodenectomy) and OPD(Open Pancreaticoduodenectomy)
Acronym: TDCBLAP
Status: Enrolling by invitation | Type: Observational
Sponsor: Zhijun Bao (Other)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Sponsor-Investigator, Zhijun Bao, Dean, Fudan University
Organization: Fudan University (Other)
Other Study IDs: SHDC2024CRI080
Record Dates: First submitted 2024-11-10; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Pancreatic Neoplasms
Keywords: pancreatic cancer; LPD; OPD; complication
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Pathological tissue,blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OPD: The patients who received the OPD
  Interventions: Procedure: LPD

INTERVENTIONS:
Procedure: LPD — The patients who received the LPD

SUMMARY:
Main objective: This project intends to design a simulated RCT project and clinically relevant RCT study to target, selecting the study titled "Short-Term outcomes Following Laparoscopic vs Open Pancreaticoduodenectomy in Patients With Pancreatic Ductal Adenocarcinoma: A Randomized Clinical Trial (Short-term Outcomes of Laparoscopic versus Open Pancreaticoduodenectomy in Patients with Pancreatic Ductal Adenocarcinoma)", use the cases in the Pancreatic Cancer Special Disease Cohort Database, compare the differences in complications and short-term prognosis between patients with pancreatic cancer after laparoscopic and open pancreaticoduodenectomy, investigate the efficacy and safety of laparoscopic pancreaticoduodenectomy, and provide the basis and reference of real-world data for clinical relevant studies. Secondary objective: To predict the incidence of postoperative complications and short-term outcomes of pancreatic cancer patients by comparing the difference of complications and short-term prognosis between laparoscopic and open pancreaticoduodenectomy, and to improve the treatment power of patients scheduled for surgery and postoperative patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years old, with no gender limit;
* Histologically confirmed or clinically diagnosed as pancreatic cancer by MDT (multidisciplinary team), without histopathological evidence;
* Patients may receive LPD or OPD according to the MDT evaluation;
* Patients understand and are willing to comply with the trial;
* Signed written informed consent before patient enrollment;
* Patients who meet the clinical guidelines for intent to treat.
* Those who met each of the above criteria were included in the study.

Exclusion Criteria:

* Patients with distant metastasis found before or during surgery, including peritoneal, liver, distant lymph node metastasis, and other organ involvement;
* Patients who need pancreatic neck or pancreatic tail, total pancreatic resection or other palliative surgery;
* Preoperative anesthesia ASA score of 4 points;
* A history of other malignant tumors;
* Pregnant or lactating women;
* Patients with severe mental disorders;
* MDT evaluates patients with vascular invasion and requiring vascular resection based on abdominal imaging data;
* Patients who have participated in other clinical trials within 3 months. Those who meet any of the above criteria were not included in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated with LPD or OPD for pancreatic cancer in Huadong Hospital from 1,January 2020 to 31,December 2022
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall survive | from the day after surgery to 3 years
complication | during the days Postoperative up to 1 year
  any possible symptoms caused by surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Huadong Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided